CLINICAL TRIAL: NCT03958617
Title: Thalamic Deep Brain Stimulation for Tourette's Syndrome: a Pragmatic Trial With Brief Randomized, Double-blinded Sham Controlled Sequences
Brief Title: Thalamic Deep Brain Stimulation for Tourette Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Jens Kuhn, P.I., University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1648
Record Dates: First submitted 2017-06-26; First posted 2019-05-22 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: A pragmatic trial with brief randomized, double-blinded sham controlled sequences
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On condition (Active Comparator): Ongoing thalamic deep brain stimulation
  Interventions: Device: Bilateral Deep brain stimulation of the thalamus, Medtronic Device
- Off condition (Sham Comparator): Switched off thalamic deep brain stimulation, sham stimulation
  Interventions: Device: Bilateral Deep brain stimulation of the thalamus, Medtronic Device

INTERVENTIONS:
Device: Bilateral Deep brain stimulation of the thalamus, Medtronic Device

SUMMARY:
In this single-center trial, we aim to include 8 patients with severe and medically refractory Tourette's syndrome. All patients undergo deep brain stimulation surgery with two electrodes located in the centromedian-parafascicular complex. Tic severity and secondary outcome measurements are assessed six and twelve months after surgery. Additionally, a short randomized, double-blinded sham controlled crossover sequence of 24 to 48 hours in either active or sham stimulation is implemented after both 6 and 12 months assesments. Subjects and clinicians are blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Das Tourette-Syndrom (ICD-10: F 95.2; DSM IV: 307.23) als Hauptdiagnose. Bei dem Patienten ist aufgrund einer chronischen, schwergradigen und therapieresistenten Verlaufsform des TS eine Behandlung mittels THS thalamischer Strukturen im Sinne einer ultima ratio vorgesehen.
* Alter des Patienten 18 bis 65 Jahre
* Sicher im Verstehen der deutschen Sprache
* Unterzeichnete Einverständniserklärung

Exclusion Criteria:

* Klinisch manifeste Psychose
* Schwangerschaft und Stillzeit
* Unterbringung nach PsychKG
* Kontraindikationen einer MRT-Untersuchung wie z. B. implantierter Herzschrittmacher / Defibrillator
* Neoplastische neurologische Erkrankungen
* Kontraindikationen einer stereotaktischen Operation, wie z. B.: erhöhte Blutungsneigung, cerebrovaskuläre Erkrankungen (z. B. arteriovenöse Malformationen, Aneurysmata, systemische Gefäßerkrankungen, die auf das Cerebrum übergreifen).
* Teilnahme an einer anderen klinischen Studie
* Hirnassoziierte Kriterien, die eine OP ausschließen (Gefäßanomalien, große arteriovenöse Malformationen, Hirnmetastasen, Neoplasien des ZNS (Ausnahme asymptomatisches inzidentielles Meningeom))
* Antikoagulationtherapie, die in der perioperativen Phase nicht ausgesetzt werden kann
* OP am Gehirn in der Anamnese, die mit der Platzierung/Funktion des MP interferieren
* Med. Gegebenheiten, die mit der Studienprozedur interferieren oder Evaluation der Studienparameter beeinträchtigen inkl. Erkrankungen im terminalen Stadium (Lebenserwartung < 12 Monate)
* Akute Suizidalität
* Abhängigkeit von Alkohol oder Drogen (exklusive Cannabis, da es von schwer betroffenen Patienten teilweise zur Ticreduktion im Sinne einer Selbstmedikation eingesetzt wird sowie exklusive Opioide und Benzodiazepine, wenn diese initial zur Ticreduktion im Sinne einer Selbstmedikation eingesetzt wurden)
* Klinisch relevante internistische oder neurologische Erkrankungen
* Intelligenzminderung
* Alle aktiv implantierten Medizinprodukte
* Schweres Schädel-Hirn-Trauma in der Anamnese
* Metallimplantate im Kopfbereich ( Bsp. Aneurysmaclips)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Change in the YGTSS Scale from Baseline to 6 and 12 months
  Motor tic subscore range 0-25 Vocal tic scubscore range 0-25 Impairment range0-50 Total Score (Vocal tic score + Motor tic score + Impairment) range 0-100
  Higher Scores indicate higher tic severity, thus worse outcome

SECONDARY OUTCOMES:
Modified Rush video rating scale (MRVRS) | Change in the MRVRS Scale from Baseline to 6 and 12 months
  Range 0-20
  Higher Scores indicate higher tic severity, thus worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kuhn, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No